CLINICAL TRIAL: NCT00290641
Title: A Cyclophosphamide/Fludarabine/Total Body Irradiation Preparative Regimen for Patients With Hematological Malignancy Receiving Unrelated Donor Umbilical Cord Blood Transplantation
Brief Title: Chemotherapy and Total-Body Irradiation Followed by Donor Umbilical Cord Blood Transplant, Cyclosporine, and Mycophenolate Mofetil in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 2000LS068; MT2000-25 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood acute myeloid leukemia in remission; secondary acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; refractory anemia with excess blasts; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; noncontiguous stage II adult Burkitt lymphoma; recurrent adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; recurrent adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; refractory anemia with excess blasts in transformation; refractory cytopenia with multilineage dysplasia; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; noncontiguous stage II adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; blastic phase chronic myelogenous leukemia; chronic idiopathic myelofibrosis; chronic eosinophilic leukemia; chronic neutrophilic leukemia; contiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; stage I adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; contiguous stage II grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent adult lymphoblastic lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory, with Excess of Blasts; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Dendritic Cell Sarcoma, Interdigitating; Leukemia, Myeloid, Acute; Lymphoma, Large-Cell, Immunoblastic; Blast Crisis; Primary Myelofibrosis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic | interventions — Filgrastim; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Biological: graft-versus-tumor induction therapy
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: umbilical cord blood transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as cyclophosphamide and fludarabine, and radiation therapy before a donor umbilical cord blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well giving chemotherapy together with total-body irradiation followed by donor umbilical cord blood transplant, cyclosporine, and mycophenolate mofetil works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the engraftment potential of unrelated allogeneic umbilical cord blood (UCB) using nonmyeloablative conditioning comprising fludarabine, cyclophosphamide, and total-body irradiation followed by post-transplant immunosuppression comprising cyclosporine and mycophenolate mofetil in patients with hematologic malignancies.

Secondary

* Determine the rate of neutrophil and platelet recovery and the completeness of donor cell engraftment in patients treated with this regimen.
* Determine the incidence and severity of acute and chronic graft-versus-host disease (GVHD) in patients treated with this regimen.
* Determine the incidence of malignant relapse in patients treated with this regimen.
* Determine the 1- and 2-year survival and event-free survival of patients treated with this regimen.
* Determine the phenotype and function of immune cells recovering after UCB transplantation in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients are stratified according to HLA disparity (0-1 vs 2) and number of graft units (1 vs 2).

* Nonmyeloablative conditioning: Patients receive nonmyeloablative conditioning comprising fludarabine IV over 1 hour on days -8 to -6 and cyclophosphamide IV over 2 hours on days -7 and -6. Patients undergo total-body irradiation twice daily on days -4 to -1.
* Unrelated allogeneic umbilical cord blood transplantation (UCBT): Patients undergo 1 or 2 unrelated allogeneic UCBTs on day 0.
* Immunosuppression: Patients receive cyclosporine orally or IV over 2 hours 2-3 times daily beginning on day -3 and continuing until day 100, followed by a taper in the absence of graft-vs-host disease (GVHD). Patients also receive mycophenolate mofetil orally or IV twice daily on days -3 to 30, continuing beyond day 30 if no donor engraftment. Patients also receive filgrastim (G-CSF) IV or subcutaneously beginning on day 1 and continuing until blood counts recover.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a hematologic malignancy of 1 of the following types:

  * Acute myeloid leukemia (AML), meeting the following criteria:

    * In complete remission (CR) by morphology (< 5% blasts in the bone marrow), as defined by 1 of the following:

      * In first CR (CR1) and meets ≥ 1 of the following high-risk criteria:

        * High-risk cytogenetics (e.g., those associated with myelodysplastic syndromes [MDS] or complex karotype)
        * Preceding MDS
        * More than 2 courses of therapy was required to obtain CR
      * In second or greater CR
    * No morphologic relapse

      * Cytogenetic relapse or persistent disease allowed
  * Acute lymphocytic leukemia (ALL), meeting the following criteria:

    * In CR, as defined by 1 of the following:

      * In CR1 and meets ≥ 1 of the following high-risk criteria:

        * Unfavorable high-risk cytogenetics [t(9;22), t(1;19), t(4;11) or other MLL rearrangements]
        * More than 1 course of therapy was required to obtain CR
      * In second or greater CR
    * No morphologic relapse or persistent disease
  * Chronic myelogenous leukemia (CML), excluding refractory blast crisis
  * Advanced myelofibrosis
  * Advanced myelodysplasia (blasts < 10% [otherwise need AML induction pre-transplant]), meeting ≥ 1 of the following criteria:

    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
    * Refractory anemia with severe pancytopenia
    * High-risk cytogenetics
  * Non-Hodgkin's lymphoma (NHL), meeting the following criteria:

    * One of the following histologic subtypes:

      * Mantle cell NHL

        * Disease progression after initial therapy (e.g., CHOP)
        * Beyond CR1 or beyond first partial remission (PR)
      * Intermediate-grade NHL in second or greater CR or PR
      * High-grade NHL

        * Stage III or IV disease AND received initial therapy
        * Stage I or II disease at diagnosis that subsequently progressed after a prior response duration of < 1 year
    * No chemotherapy-refractory NHL (i.e., < progressive disease after > 2 salvage regimens)
* Donor available, meeting the following criteria:

  * No other existing HLA-identical related donor available
  * 4-6/6 HLA-A, -B, and -DRB1, matched unrelated donor by molecular techniques

    * A and B to antigen level resolution
    * DR to allele resolution
  * Umbilical cord blood (UCB) graft may consist of one or two UCB units NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* Karnofsky score 80-100% (for adults) OR
* Lansky score 50-100% (for children)
* Creatinine ≤ 2.0 mg/dL (for adults) OR creatinine clearance > 40 mL/min (for children)

  * Adults with a creatinine > 1.2 mg/dL or a history of renal dysfunction must have a creatinine clearance > 40 mL/min
* Bilirubin ≤ 2 times normal
* AST and ALT ≤ 2 times normal
* Alkaline phosphatase ≤ 2 times normal
* Pulmonary function > 50 % of normal
* LVEF ≥ 45%
* No active infection, including Aspergillus or other mold, within the past 30 days
* No history of HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior myeloablative transplant within the past 6 months if ≤ 18 years old
* No prior myeloablative allotransplant or autologous transplant if > 18 years old
* No prior extensive therapy (e.g., > 12 months of alkylating therapy or > 6 months of alkylating therapy with extensive radiation)

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2001-04; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Engraftment as measured by an absolute neutrophil count of donor origin > 0.5 x 109 /L for 3 days by day 42

SECONDARY OUTCOMES:
Incidence and severity of acute or chronic graft-versus-host-disease, relapse, or mortality at day 100
Survival and event-free survival by Kaplan-Meier estimation at 1 and 2 years after umbilical cord blood (UCB) transplant

CONTACTS AND LOCATIONS:
Overall Officials: Claudio G. Brunstein, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Barker JN, Weisdorf DJ, DeFor TE, Blazar BR, McGlave PB, Miller JS, Verfaillie CM, Wagner JE. Transplantation of 2 partially HLA-matched umbilical cord blood units to enhance engraftment in adults with hematologic malignancy. Blood. 2005 Feb 1;105(3):1343-7. doi: 10.1182/blood-2004-07-2717. Epub 2004 Oct 5. PMID 15466923